CLINICAL TRIAL: NCT03160625
Title: Evaluation of Rate Adaptive Pacing on Chronotropic Response in Preserved Ejection Fraction HF
Acronym: RESPOND-HF
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of eligible patient.
Sponsor: Medtronic Cardiac Rhythm and Heart Failure (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: RESPOND-HF
Record Dates: First submitted 2017-03-22; First posted 2017-05-19 (Actual); Last update posted 2018-04-19 (Actual); Status verified 2018-04

CONDITIONS: Heart Failure With Preserved Ejection Fraction

STUDY DESIGN:
Intervention Model Description: To assess whether rate adaptive pacing provides benefit to HFpEF patients, a pool of up to 60 qualifying subjects with pre-existing pacemaker and established diagnosis of HFpEF who demonstrate chronotropic incompetence (CI) with RAP turned off will be enrolled.
  Subjects who meet CI criterion during Visit 2 will be randomized. Subjects' principal investigator and study team will be blinded to the randomization assignment. However clinical site personnel performing the device programming will not be blinded. Site personnel performing the CPET and 6-min hall walk assessments will be blinded to the randomization assignment.
  Crossover of study subjects will occur during Visit 3, which will occur 12 weeks after subject enrollment. Subjects who were randomized with RAP ON first will have the device programmed to RAP OFF and conversely, subjects who were randomized to RAP OFF first will have the device programmed to RAP ON.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Subjects' principal investigator and study team will be blinded to the randomization assignment. However clinical site personnel performing the device programming will not be blinded. Site personnel performing the CPET and 6-min hall walk assessments will be blinded to the randomization assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Rate Adaptive Pacing ON (Active Comparator): The Rate Adaptive Pacing (RAP) feature in the Medtronic implantable pulse generator (IPG) will be programmed to level 4 (More Active Lifestyle) with ADL rate of 95 bpm or higher, and Upper sensor rate that is subject's age predicted maximum heart rate. The age predicted maximum heart rate (APMHR) will be computed as: APHMR = 220 - age
  Interventions: Device: Rate Adaptive Pacing
- Rate Adaptive Pacing OFF (Active Comparator): The Rate Adaptive Pacing (RAP) feature in the Medtronic implantable pulse generator (IPG) will be turned off for this arm of the study.
  Interventions: Device: Rate Adaptive Pacing

INTERVENTIONS:
Device: Rate Adaptive Pacing — Rate Adaptive Pacing varies the pacing rate in response to the patient's physical motion as detected by an activity sensor.

SUMMARY:
RESPOND-HF is a prospective, multi-center, non-significant risk pilot study with cross-over design. The purpose of the study is to investigate if rate adaptive pacing has the potential to provide benefit to HF patients with preserved ejection fraction, referred to as HFpEF patients. Findings from this pilot study may be used to guide subsequent efforts to design and conduct a prospective, randomized, multi-center pivotal trial powered to show improvement in patient outcomes.

DETAILED DESCRIPTION:
The RESPOND-HF is a prospective, multi-center, investigational, pilot study with cross-over design. Patients with existing pacemakers who have been diagnosed with HFpEF and meet study inclusion/exclusion criteria will be included in the study.

The study is expected to be conducted at up to 5 centers in the United States and up to 300 patients will be consented to enroll up to 100 qualifying patients . Up to 60 patients meeting chronotropic incompetence (CI) criterion will be enrolled. The study will be conducted in subjects who have previously (≥ 30 days) been implanted with Medtronic, dual chamber pacemaker (IPG) device with rate adaptive pacing (RAP) feature. Additionally, up to 40 patients who do not meet CI criterion will be enrolled to collect ambulatory activity and heart rate data using AVIVO/SEEQ patch. These patients will be followed for only 1 week. It is estimated that subject enrollment will take approximately 12 to 18 months, with a study follow-up of 18 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years or legal age to provide informed consent
* Willing and be able to provide informed consent
* Previous clinical diagnosis of HF and exhibits HF signs and symptoms consistent with NYHA II or III (or class B or C)
* Chronic Rx for heart failure with loop diuretic or a mineralocorticoid receptor antagonist (MRA)
* LVEF ≥ 45% within previous 12 months. Acceptable methods include echo, ventriculogram (angiography or nuclear), nuclear stress test. If patient has a prior history of significant left ventricular systolic dysfunction defined as EF < 0.40, patient must have a HF event within previous 12 months defined as:

  * Hospitalization for decompensated HF
  * Unscheduled treatment for HF with intravenous loop diuretic or hemofiltration
* On stable HF medical therapy for previous 30 days. Dose changes of ACEI / ARB and beta blockers of less than 50% increase or decrease are acceptable for stability
* Treadmill exercise time using modified Naughton protocol of greater than 3 min and less than 15 min for men and 14 for women
* Medtronic dual chamber pacemaker implanted for ≥ 30 days
* Sinus rhythm at rest

Exclusion Criteria:

* Women who are pregnant or plan to become pregnant
* Life expectancy less than 1 year
* Enrollment in any concurrent study that could potentially be confounding
* Orthopedic, neuromuscular or any other condition limiting exercise testing
* Unstable angina or MI or have undergone CABG/PTCA within previous 60 days
* A candidate for CABG/PTCA at the time of informed consent
* Use of inotrope therapy on a regular basis (e.g. daily, weekly etc.)
* Severe and/or poorly controlled major active comorbidity, including (but not limited to):

  * Diabetes: Hb1AC > 9.5
  * Severe COPD: e.g. end stage emphysema managed using 2 or more inhalers and/or using home oxygen
  * Severe pulmonary disease limiting functional capacity
  * Hypertension: SBP > 160 mmHg at time of screening
  * Cancer: Ongoing therapy or therapy within previous 3 months
  * Severe valvular disease
  * Renal impairment with serum creatinine > 3 mg/dL
  * Anemia with hemoglobin < 8 g/dL or major bleeding event within the past 60 days
* Primary diagnosis of pulmonary arterial hypertension with ongoing severe pulmonary hypertension and treatment
* Known familial hypertrophic cardiomyopathy or hypertrophic obstructive cardiomyopathy
* Known restrictive cardiomyopathy or systemic illness known to be associated with infiltrative myocardial disease (e.g. amyloidosis, sarcoidosis, hemochromatosis)
* Pericardial restriction or hemodynamically significant pericardial effusion
* Patients expected to undergo device or lead replacement within study follow-up duration
* Allergies to hydrogel in SEEQ/AVIVO patch
* Patients who are expected to be ventricular paced over 40% of the time
* Long standing persistent AF Or Ongoing episode of persistent AF

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-07-01 (Estimated); Primary Completion 2018-04-30 (Estimated); Study Completion 2018-05-31 (Estimated)

PRIMARY OUTCOMES:
Exercise time | 18 Weeks
  Exercise time on a treadmill guided by respiratory exchange ratio (RER) during cardiopulmonary exercise test (CPET).

SECONDARY OUTCOMES:
Peak VO2 | 18 Weeks
  Maximum rate of oxygen consumption during treadmill testing
Peak metabolic equivalents (METs) | 18 Weeks
  Ratio of the rate of energy expended during treadmill testing to the rate of energy expended at rest
Peak respiratory exchange ratio (RER) | 18 Weeks
  Maximum ratio between the amount of carbon dioxide (CO2) produced and oxygen (O2) used during treadmill testing
VE/VO2 slope | 18 Weeks
  Minute ventilation oxygen consumption relationship
VO2 at Ventilator Anaerobic Threshold (VAT) | 18 Weeks
  Rate of oxygen consumption at VAT during treadmill testing
VCO2 at Ventilator Anaerobic Threshold (VAT) | 18 Weeks
  Rate of carbon dioxide production at VAT during treadmill testing
KCCQ | 18 Weeks
  Subject's quality of life measure using KCCQ
6 Minute Hall Walk | 18 Weeks
  Subject's activity of daily living as measure by 6 minute hall walk
Daily Activity | 18 Weeks
  Activity data collected by the implantable device and wearable sensor (SEEQ/AVIVO patch)
Global Patient Health Assessment | 18 Weeks
  Global patient health status using 0-100 visual analog scale
NT-proBNP | 18 Weeks
  N-terminus pro Brain Natriuretic Peptide
Correlation between activity and HR | 18 Weeks
  Correlation between activity and heart rate

CONTACTS AND LOCATIONS:
Overall Officials: Aida Cicic, MD, Study Director — Medtronic
Locations (5):
- United States (5):
  - Mayo Clinic (Rochester MN), Rochester, Minnesota
  - Mid America Heart Institute (MAHI), Kansas City, Missouri
  - Lindner Research Center, Cincinnati, Ohio
  - Ohio State University, Columbus, Ohio
  - Lancaster General Hospital, Lancaster, Pennsylvania

IPD SHARING:
Plan to Share IPD: No